CLINICAL TRIAL: NCT01575158
Title: Citalopram vs Clomipramine vs Placebo in Recurrent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish University Antidepressant Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUAG-5
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Citalopram; Clomipramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- citalopram (Experimental): citalopram
  Interventions: Drug: Citalopram
- clomipramnine (Active Comparator): clomipramine
  Interventions: Drug: Clomipramine
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Citalopram
  Arms: citalopram
Drug: Clomipramine
  Arms: clomipramnine
Drug: placebo
  Arms: placebo

SUMMARY:
citalopram and clomipramine are better than placebo in preventing new episodes of depression in patients with recurrent depression

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent depression
* Sustained response achieved (3 consecutive monthly ratings at the HDS below 13)after a treatment requiring index episode

Exclusion Criteria:

* Contraindications to study medications
* Pregnancy
* Substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1997-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
2 Hamilton Depression Rating Scale scores of at least 16 with one weeks interval or initiation of another antidepressant treatment | 2 years of follow-up

SECONDARY OUTCOMES:
Study termination due to adverse event or non-compliance | 2 years of follow-up